CLINICAL TRIAL: NCT04570241
Title: Evaluation of the Effect of Mobilization at School Level on Behaviour Change in Favor of Malaria Control in the Health District of Mbandjock in Cameroon
Brief Title: Mobilization at the Level of Schools on the Behavioral Change in Favor of the Fight Against Malaria in Mbandjock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cameroon Coalition Against Malaria (CCAM) (Other)
Responsible Party: Principal Investigator, Pr Wilfred Fon Mbacham, Principal Investigator, Cameroon Coalition Against Malaria (CCAM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCCCAM/10/02/2016
Record Dates: First submitted 2020-09-14; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Malaria
Keywords: Malaria; Awareness; Knowledge; Attitudes; Practices
MeSH Terms: conditions — Malaria; Behavior

STUDY DESIGN:
Intervention Model Description: A 2-arm, open-label, randomized controlled clinical trial will be adopted with the Mbandjock health district as the test district and Sa'a Health District a Control Health District.
  The Lot Quality Assurance Sampling (LQAS) method was used. Since this method requires that the intervention zones be divided into supervision areas, the health areas of each district were considered as supervision areas. The health area was selected in the ratio 2:1. In the test district 11 health areas were used and 6 health district in the control district. 19 households were selected for each health area as required by the LQAS method.
  A total of 209 pupils and 209 adults shall be enrolled from households in Mbandjock. Similarly, 114 pupils and 114 adults will be recruited in Sa'a. In addition, 57 teachers shall be enrolled in the District of Mbandjock only. A total of 703 participants shall be enrolled during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A-Malaria toolkit (Active Comparator): School children shall be trained on key malaria messages with a malaria toolkit. From the training received, the pupils will carry out awareness-raising in communities with key messages learnt.
  Interventions: Behavioral: Malaria toolkit
- Group B-No malaria toolkit (No Intervention): School children shall not be trained on key malaria messages with a malaria toolkit. Pupils will not carry out awareness-raising in communities with key messages.
  .

INTERVENTIONS:
Behavioral: Malaria toolkit — Knowledge, attitude, and practice on malaria
  Arms: Group A-Malaria toolkit

SUMMARY:
The main aim of this study is to determine the effect of awareness campaigns by school children targeting their communities on knowledge, attitudes, and practices in malaria control in the Mbandjock health district. A two-arm, open-label, randomized controlled clinical trial will be adopted with the Mbandjock Health District as the test district and Sa'a Health District as control Health District. This will last from January 2017 to December 2020. The Lot Quality Assurance Sampling (LQAS) method was used. The health area was selected in the ratio 2:1. A total of 209 pupils and 209 adults shall be enrolled from households located in Mbandjock. Similarly, 114 pupils and 114 adults will be recruited in Sa'a. In addition, 57 teachers shall be enrolled in the District of Mbandjock only. A total of 703 participants shall be enrolled during the study.

DETAILED DESCRIPTION:
General objective To determine the effect of awareness campaigns by school children targeting their communities on knowledge, attitudes and practices in malaria control in the Mbandjock health district.

Specific objectives

* To describe the socio-demographic characteristics of households in the health districts of Mbandjock and Sa'a at the time of the survey;
* To measure the change due the intervention on knowledge of malaria transmission, diagnosis, treatment and prevention in the health district of Mbandjock;
* To measure the change due the intervention on attitudes towards malaria diagnosis, treatment and prevention in the Mbandjock health district;
* To measure the change due the intervention on practices in the diagnosis, treatment and prevention of malaria in the Mbandjock health district.

Methodology Study design A two-arm, open label, randomized controlled clinical trial will be adopted with Mbandjock health district as the test district and Sa'a Health District a Control Health District.

Study site and study population The study population will be the entire population of the Mbandjock and Sa'a communities.

Sampling method The Lot Quality Assurance Sampling (LQAS) method was used. Since this method requires that the intervention zones be divided into supervision areas, the health areas of each district were considered as supervision areas. The health area was selected in the ratio 2:1. In the test district 11 health areas were used and 6 health district in the control district. 19 households were selected for each health area as required by the LQAS method.

Sample size A total of 209 pupils and 209 adults shall be enrolled from households in Mbandjock. Similarly, 114 pupils and 114 adults will be recruited in Sa'a. In addition, 57 teachers shall be enrolled in the District of Mbandjock only. A total of 703 participants shall be enrolled during the study.

Duration of study The study duration is three years. This will last from January 2017 to December 2020.

ELIGIBILITY:
Inclusion Criteria:

* Children should be of school-going age.
* Children belong to an authorized school.
* Adult belonging to a household.

Exclusion Criteria:

* Children not going to school.
* Children not belonging to an authorized school.
* An adult that cannot be identified with any household.

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 703 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of school children to be trained with the malaria toolkit in order to educate adults on malaria control in different communities in the Mbandjock Health District | 24 months
  The intervention group will include 209 children to be trained with a toolkit on malaria in order to educate 209 adults in their different communities

CONTACTS AND LOCATIONS:
Overall Officials: Esther Talla, MD, Study Director — MC-CCAM
Locations (1):
- Mbandjock Health District, Yaoundé, Centre Region, Cameroon

IPD SHARING:
Plan to Share IPD: Yes
Data on knowledge, attitude, and practice of malaria will be shared with the scientific community and policy makers
Supporting Information: CSR
Time Frame: December 2020 and for a period of at least 10 years
Access Criteria: Must be a researcher or policy marker